CLINICAL TRIAL: NCT05434247
Title: A Prospective Randomized Study Comparing the Diagnostic Adequacy of 25-gauge Fork-tip, Franseen and Reverse-bevel Type Needles in Endoscopic Ultrasound Guided Tissue Acquisition
Brief Title: Comparing the Diagnostic Adequacy of 25-gauge Fork-tip, Franseen and Reverse-bevel Type Needles in Endoscopic Ultrasound Guided Tissue Acquisition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Alexandra Hospital, Brisbane, Australia (Other)
Responsible Party: Principal Investigator, Alexander Huelsen, Gastroenterology Staff Specialist, Princess Alexandra Hospital, Brisbane, Australia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LNR/QMS/44303
Record Dates: First submitted 2022-03-19; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Biopsy, Needle
Keywords: Endoscopic ultrasound, Fine Needle Biopsy

STUDY DESIGN:
Intervention Model Description: Randomized trial with retrospective comparator group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Reverse-bevel ProCore™ (Other): Historical comparator group of biopsies taken using Echo Tip® HD ProCore™ (Wilson-Cook Medical Inc., Winston-Salem, NC, United States) biopsy needle. Slow pull stylet technique with rapid on site evaluation in all cases.
  Interventions: Device: Needle choice
- Fork-tip SharkCore™ (Experimental): Experimental group of biopsies using SharkCore™ (Medtronic Inc., Sunnyvale, CA, United States) biopsy needle. Slow pull stylet technique with rapid on site evaluation in all cases.
  Interventions: Device: Needle choice
- Franseen Acquire™ (Experimental): Experimental group of biopsies using Acquire™ (Boston Scientific, Marlborough, MA, United States) biopsy needle. Slow pull stylet technique with rapid on site evaluation in all cases.
  Interventions: Device: Needle choice

INTERVENTIONS:
Device: Needle choice — The type of needle use was the only intervention

SUMMARY:
Endoscopic ultrasound guided fine needle aspiration (EUS-FNA) and fine needle biopsy (EUS-FNB) are well established techniques for the acquisition of tissue to classify a number of lesions of the gastrointestinal tract and surrounding organs. These include pancreatic, lymphoid, subepithelial and other abdominal lesions. Historically, FNA was the sole available modality used to obtain cytological samples for analysis. The major shortcoming of this technique is the lack of a histological tissue core.

In recent years attention has turned to optimizing needle design to improve sample quality. New needles have been developed which aim to obtain a core of tissue with preserved architecture.

These needles include the first generation Reverse-bevel Echo Tip® HD ProCore™ (Wilson-Cook Medical Inc., Winston-Salem, NC, United States), and the second generation Fork-tip SharkCore™ (Medtronic Inc., Sunnyvale, CA, United States) and Franseen Acquire™ (Boston Scientific, Marlborough, MA, United States).

Currently there are a paucity of studies comparing the performance of these needles, and only two of these are prospective randomized controlled trials. Real world performance of these needles has seldom been reported, with only one RCT including non-pancreatic masses in their analysis.

The investigators hypothesize that second generation needles have equivalent or better diagnostic performance than the prior first-generation needle.

To test this, the investigators aim to conduct a prospective randomized controlled study comparing the performance of Fork-tip and Franseen needles for the sampling of pancreatic, subepithelial, lymphoid and other abdominal or mediastinal lesions. They also aim to include a retrospective control arm of consecutive cases using the first-generation Reverse-bevel needle.

The investigatora aim to assess the diagnostic yield of each needle, as well as number of needle passes used, and specimen quality.

ELIGIBILITY:
Inclusion Criteria:

* Any solid tissue biopsy performed at the time of endoscopic ultrasound

Exclusion Criteria:

* Fluid samples were excluded.
* Cases where biopsy was not deemed necessary by the proceduralist based on endosonographic findings
* Cases where biopsy was deemed unsafe

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | At study completion, approximately 1 year after final subject enrolled
  The percentage of lesions sampled for which a tissue diagnosis was obtained

SECONDARY OUTCOMES:
Number of needle passes | At study completion, approximately 1 year after final subject enrolled
Sample bloodiness | At study completion, approximately 1 year after final subject enrolled
  A subjective assessment of the amount of blood seen on histopathological specimens (1 = no interference with interpretation, 2 = interference with interpretation but diagnosis can still be made, 3 = excessive blood makes assessment impossible)
Target tissue cellularity | At study completion, approximately 1 year after final subject enrolled
  Subjective assessment by histopathologist of the cellularity of the sample (consisting of cells from the target lesion) - low, medium or high.

OTHER OUTCOMES:
Adverse events | At end of study medical record review, approximately 1 year after final subject enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Huelsen, MD, Study Director — QLD Health
Locations (1):
- Princess Alexandra Hospital, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No